CLINICAL TRIAL: NCT00349973
Title: Clinical Trial of Dipyridamole in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, L. Elliot Hong, Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HP-00043347
Record Dates: First submitted 2006-07-05; First posted 2006-07-10 (Estimated); Results first posted 2018-12-10 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder
Keywords: Schizophrenia; Positive symptoms; Negative symptoms; Cognitive deficits
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Cognition Disorders | interventions — Dipyridamole; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Dipyridamole
  Interventions: Drug: Dipyridamole
- 2 (Active Comparator): Olanzapine
  Interventions: Other: Olanzapine

INTERVENTIONS:
Drug: Dipyridamole — Week 1- 50 mg bid Week 2- 50 mg am and 100 mg pm Weeks 3-6 100 mg am and 100 mg pm
  Arms: 1
Other: Olanzapine — Week 1- 5 mg BID Week 2- 5 mg am and 10 mg pm Weeks 3-6 10 mg am and 10 mg pm
  Arms: 2

SUMMARY:
This is a 6-week, randomized, double blind, parallel groups designed, olanzapine-controlled trial of oral dipyridamole in symptomatic patients with a (DSM IV) diagnosis of schizophrenia, schizoaffective or schizophreniform disorder. This pilot study aims to provide preliminary estimates of whether the effect sizes of dipyridamole on positive symptoms, negative symptoms, and cognitive deficits differ between schizophrenia patients treated with dipyridamole, and schizophrenia patients treated with olanzapine. A total of 30 subjects will be recruited locally.

DETAILED DESCRIPTION:
Since the demonstrated success of chlorpromazine in treating psychosis in the1950's, the pharmacotherapy of schizophrenia has focused mainly on drugs with antidopaminergic actions. These drugs have robust effects on reality distortion and disorganization symptom complexes, but minimal effect on cognitive impairment, negative symptoms, and functional outcome and quality of life measures. Newer generation antipsychotic drugs have a similar profile of effects, with some advantages on the course of depression, hostility, suicide, hospital readmission rates and motor side effect measures. Side effects such as weight gain, increase in cardiovascular stress and diabetes risk are associated with some new generation drugs. A new class of drugs is needed to address the inadequate effectiveness and the side-effect disadvantages of the currently available pharmacological agents for the treatment of schizophrenia. Recently, new treatment strategies using nicotinergic drugs or agonists at the glycine modulatory site of the glutamatergic N-methyl-D-aspartate (NMDA) receptor have been employed in clinical trials with mixed results. Our proposal focuses on a clinically available adenosine agonist, dipyridamole, in a 6-week clinical trial. Published data suggest effectiveness of dipyridamole in treating psychosis when added to haloperidol treatment. The effectiveness of dipyridamole alone in treating schizophrenia symptoms, although indirectly suggested by several lines of evidence, has not been tested.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between ages 18-65, both males and nonpregnant females (on birth control) Diagnosis of schizophrenia, schizoaffective or schizophreniform disorder Ability to give written informed consent Total BPRS score > 27 Psychosis subscale scores > 7

Exclusion Criteria:

* Patients with coagulative disorders, bleeding diathesis or currently on anticoagulants, and patients with major medical illnesses (including hypertension, angina, and cardiovascular diseases) or an abnormal baseline ECG.

Patients with moderate to severe mental retardation.

Inability to sign informed consent.

Patients with a history of serious violence (e.g., suicide attempts, or assaultive behavior).

Patients on clozapine treatment within the 6 weeks leading to the double-blind phase.

Patients with a history of olanzapine non-response

Positive Urine Toxicology Screen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2001-05; Primary Completion 2008-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ikwunga Wonodi, MD, Study Director — Maryland Pschiatric Research Center, University of Maryland School of Medicine; Gunvant K Thaker, MD, Principal Investigator — University of Maryland, College Park
Locations (1):
- Maryland Psychiatric Research Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Akhondzadeh S, Shasavand E, Jamilian H, Shabestari O, Kamalipour A. Dipyridamole in the treatment of schizophrenia: adenosine-dopamine receptor interactions. J Clin Pharm Ther. 2000 Apr;25(2):131-7. doi: 10.1046/j.1365-2710.2000.00273.x. PMID 10849191
- [Result] Dixon DA, Fenix LA, Kim DM, Raffa RB. Indirect modulation of dopamine D2 receptors as potential pharmacotherapy for schizophrenia: I. Adenosine agonists. Ann Pharmacother. 1999 Apr;33(4):480-8. doi: 10.1345/aph.18215. PMID 10332540
- [Result] Ferre S. Adenosine-dopamine interactions in the ventral striatum. Implications for the treatment of schizophrenia. Psychopharmacology (Berl). 1997 Sep;133(2):107-20. doi: 10.1007/s002130050380. PMID 9342776
- See also: Maryland Psychiatric Research Center — http://www.mprc.umaryland.edu/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Four participants were excluded prior to randomization (1:positive urine tox screen; 1:participant uncooperative with clinical interview; 1:withdrew consent; 1:history of cardiovascular disease).
Groups:
- Dipyridamole: Dipyridamole
  Dipyridamole : Week 1- 50 mg bid Week 2- 50 mg am and 100 mg pm Weeks 3-6 100 mg am and 100 mg pm
- Olanzapine: Olanzapine
  Olanzapine : Week 1- 5 mg BID Week 2- 5 mg am and 10 mg pm Weeks 3-6 10 mg am and 10 mg pm
Period: Overall Study
Arm/Group | Dipyridamole | Olanzapine
Started | 12 | 8
Completed | 8 | 5
Not Completed | 4 | 3
Not completed — Adverse Event | 3 | 3
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dipyridamole | Olanzapine | Total
Number analyzed (Participants) | 12 | 8 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 8 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 7 | 4 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 4 | 10
  White | 6 | 4 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Positive Symptoms by Treatment Assignment
Description: The Brief Psychiatric Rating Scale (BPRS) consists of 20 items, with 6 of these items used to assess positive symptom change. The BPRS positive symptom items are: somatic concern, conceptual disorganization, hostility, suspiciousness, hallucinatory behavior, and unusual thought content. Each scale ranges from "1=Not Present" to "7=Very Severe". A higher score indicates a more severe positive symptom rating.
Time Frame: Baseline and follow-up
Population: Participants completing the BPRS assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dipyridamole | Olanzapine
Number analyzed (Participants) | 9 | 5
units on a scale
  Baseline - Somatic Concern | 2.222 (1.716) | 1.400 (0.548)
  Follow-Up - Somatic Concern: number analyzed (Participants) | 5 | 2
  Follow-Up - Somatic Concern | 1.60 (1.34) | 1.00 (0.00)
  Baseline - Conceptual Disorganization | 2.667 (1.225) | 2.600 (0.894)
  Follow-Up - Conceptual Disorganization: number analyzed (Participants) | 5 | 2
  Follow-Up - Conceptual Disorganization | 2.00 (1.41) | 2.00 (1.41)
  Baseline - Hostility | 1.222 (0.667) | 1.200 (0.447)
  Follow-Up - Hostility: number analyzed (Participants) | 5 | 2
  Follow-Up - Hostility | 1.00 (0.00) | 2.00 (1.41)
  Baseline - Suspiciousness | 4.11 (1.54) | 3.40 (1.82)
  Follow-Up - Suspiciousness: number analyzed (Participants) | 5 | 2
  Follow-Up - Suspiciousness | 3.000 (1.581) | 1.500 (0.707)
  Baseline - Hallucination | 2.67 (2.12) | 3.80 (1.30)
  Follow-Up - Hallucination: number analyzed (Participants) | 5 | 2
  Follow-Up - Hallucination | 2.600 (2.191) | 2.500 (0.707)
  Baseline - Unusual Thought Content | 3.111 (1.167) | 3.400 (0.894)
  Follow-Up - Unusual Thought Content: number analyzed (Participants) | 5 | 2
  Follow-Up - Unusual Thought Content | 2.800 (2.168) | 1.500 (0.707)

2. Primary Outcome: Change in Negative Symptoms by Treatment Assignment
Description: The Scale for the Assessment of Negative Symptoms (SANS) total score, minus the global items, inappropriate affect, poverty of content of speech, and attention items, used to measure negative symptoms. Mean SANS total score by treatment and week. SANS total score range = 0-85. Higher scores indicate more severe negative symptoms.
Time Frame: Baseline and Follow-Up
Population: Participants completing SANS assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dipyridamole | Olanzapine
Number analyzed (Participants) | 9 | 5
units on a scale
  Baseline (Phase 1/Week 1) | 23.3 (14.7) | 25.6 (20.5)
  Follow-Up (Phase 4/Week 1): number analyzed (Participants) | 5 | 2
  Follow-Up (Phase 4/Week 1) | 25.8 (10.7) | 27.0 (29.7)

3. Primary Outcome: The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS)
Description: The RBANS is a brief, individually administered test designed to evaluate neuropsychological status of adults, ages 20-89. The 12 subtests measure attention, language, visuospatial/constructional abilities, and immediate and delayed memory. The raw scores from the subtests are scaled together to create index scores, and these are summed for conversion to a total scale score. Higher score equals a better outcome. The total index score range for the RBANS is 40-160.
Time Frame: Baseline and Follow-Up
Population: Participants completing cognitive testing.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dipyridamole | Olanzapine
Number analyzed (Participants) | 5 | 2
units on a scale
  Baseline (Phase 1/Week 1) | 73.00 (15.41) | 59.00 (1.41)
  Follow-Up (Phase 3/Week 6) | 77.40 (14.83) | 65.00 (2.83)

ADVERSE EVENTS:
Arm/Group | Dipyridamole | Olanzapine
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/8
Other Adverse Events (participants affected / at risk) | 0/12 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No